CLINICAL TRIAL: NCT06135129
Title: Diagnostic Value of SonoElastography in Evaluation of Median Nerve Changes With Rheumatoid Arthritis Patients Without Symptoms of Carpal Tunnel Syndrome
Brief Title: SonoElastography of Median Nerve in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marco Magdy Wadie, Resident doctor, Assiut University
Other Study IDs: Elastography median nerve
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Elastography
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sonoelastography — Sonoelastography (SE) is a new ultrasound-based method measure the stiffness or elasticity of tissues, has no hazards on poatients.

SUMMARY:
To assess the role of ultrasonography and SE in detecting the median nerve changes before progression to CTS in patients with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) presents with persistent pain, stiffness, progressive joint destruction, functional disability, and progressive morbidity and mortality, and is a chronic systemic autoimmune disease.1 The cause of RA remains unknown, but the pathological mechanism of synovial inflammation may result due to the complex interplay of genetic immunology and environmental factors.2 Early diagnosis is fundamental to prevent the permanent sequel of RA. Recent advances in diagnostic imaging in rheumatology have benefited patients clinically and also provided information related to the pathophysiology of diseases like arthritis.

Ultrasound (US) and magnetic resonance imaging were most commonly used in diagnosing and monitoring RA progression in joints and related joint structures.3 US elastography measures tissue elasticity using high-frequency sound waves to assess tissue's static or dynamic deformation behavior after a stimulus is applied. This technique has been described most commonly in the context of isotropic tissues, such as the liver and neoplastic diseases, but is now becoming of more interest in anisotropic tissues, such as those in the musculoskeletal system.4

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with RA and ruling out CTS by clinical evaluation that included Phalen's test, a manual muscle test of the abductor's muscle, and a search for Tinel-like signs and thenar muscle atrophy. Controls - Age- and sex- matched cases without RA undergoing US for causes unrelated to RA or CTS. The criteria for RA were adopted from The American Rheumatism Association (1987) for the classification of RA.

Exclusion Criteria:

* History of a condition other than RA that could cause CTS (e.g., diabetes mellitus, acute trauma, pregnancy ,hypothyroidism, hyperthyroidism, connective tissue disease)History of surgery for a wrist or hand fracture.
* History of other systemic neurological disorders or radiculopathy Bifid median nerve or any mass lesion identified on US examination Pregnant patients were excluded.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with RA and ruling out CTS by clinical evaluation
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
To assess the role of ultrasonography and SE in detecting the median nerve changes before progression to CTS in patients with RA. | Baseline
  The accuracy of Sonoelastography to detect median nerve changes in rheumatoid arthritis patients

REFERENCES:
- [Background] Hammer HB, Haavardsholm EA, Kvien TK. Ultrasonographic measurement of the median nerve in patients with rheumatoid arthritis without symptoms or signs of carpal tunnel syndrome. Ann Rheum Dis. 2007 Jun;66(6):825-7. doi: 10.1136/ard.2006.055988. Epub 2006 Dec 14. PMID 17170055
- [Result] Atan Uzun C, Sunar I, Gunendi Z, Gogus FN. Comparison of the median and ulnar nerves of rheumatoid arthritis patients and healthy subjects by ultrasound. Arch Rheumatol. 2022 Oct 21;38(2):183-188. doi: 10.46497/ArchRheumatol.2023.9027. eCollection 2023 Jun. PMID 37680523